CLINICAL TRIAL: NCT04651582
Title: Assessing Cognitive and Psychosocial Mechanisms of Useful Field of View Cognitive Training Using Ecological Momentary Assessment
Brief Title: The Everyday Function Intervention Trial
Acronym: EFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lesley A. Ross, Professor, Clemson University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R21AG060216 (NIH); R21AG060216 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2020-12-03 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Change; Cognitive Impairment; Healthy Aging; Dementia
Keywords: Brain training; Cognitive training; Brain health; Everyday functioning
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): 20 hours of computerized brain exercises
  Interventions: Behavioral: Cognitive Training
- Cognitively Stimulating Activities (Active Comparator): 20 hours of computerized brain exercises
  Interventions: Behavioral: Cognitive Stimulating Activities

INTERVENTIONS:
Behavioral: Cognitive Training — 20 hours of computerized activities designed to improve processing speed and divided attention
  Arms: Cognitive Training
Behavioral: Cognitive Stimulating Activities — 20 hours of traditional computer games
  Arms: Cognitively Stimulating Activities

SUMMARY:
Loss of independence, cognitive decline, and difficulties in everyday function are areas of great concern for older adults and their families. From a public health perspective, successful efforts that enable older adults to age within their homes, as compared to nursing homes, will save an estimated $80 billion dollars per year. Cognitive training is one intervention that maintains cognition, everyday function, and health. Although clearly an important and effective intervention, the mediators, or mechanisms, underlying this program are unknown. Our overall objective is to assess the cognitive and psychosocial factors within daily life that account for the transfer of one form of cognitive training to everyday function. This exploratory double-blind trial will randomize older adults to 20 hours of cognitive training or cognitively stimulating activities. The investigators will assess cognitive and psychosocial factors before, during, and after training within daily life. The investigators will then compare such factors and assess how they impact the transfer of cognitive training to everyday functioning. The investigators will also include an eligible sub group of the EFIT participants who will have functional MRI brain scans and sleep evaluation using the Sleep Profiler, a clinically approved device, at pre and post brain training. The investigators will also monitor daily activity in this sub group using FitBIt watches.

Our central hypothesis is that improvements in daily processing speed and attention, key components of higher order cognitive functions, will have the strongest relationship with everyday function changes. This exploratory study is the first of its kind and will be used to provide important data relevant to a future larger randomized controlled trial examining mediators of cognitive training in a representative sample of adults. Additionally, all data collection, with the exception of MRI, can be completed remotely within the participant's home. This information will assist in the future development of more effective home- and community-based interventions that maintain everyday function.

DETAILED DESCRIPTION:
The EFIT study is a randomized clinical trial to explore moderators and mechanisms underlying the transfer of one cognitive training program to maintained cognition and everyday function. 100 participants will complete three traditional assessments of cognitive, psychosocial, and lifestyle assessments on a study-provided laptop at baseline, post-test, and three-month follow-up. Across this study period, participants will complete daily cognitive, psychosocial, and health assessments using a study-provided smartphone. Between baseline and post-test, participants will be randomized to one of two arms: cognitive training or an active control. Both groups will complete 20 hours of activities on the study-provided laptop across a ten week period.

A subsample of 40 participants will also complete three additional measures. First, they will be provided a FitBit and be asked to wear the FitBit across the study period. Second, sleep measures will be obtained across two nights at baseline and post-test using an at home sleep monitor, which is clinically approved, and evaluated by a physician specializing in sleep. Finally, this subsample will also complete a fMRI session at baseline and posttest.

Except for the fMRI sessions, all data collection is complete remotely within the participants' homes.

ELIGIBILITY:
* Community-dwelling adults aged 65 to 90
* Ability to understand and communicate with written and spoken English
* No reported diagnosis or evidence of Alzheimer 's disease or other dementia; score of 5 or greater on the MIS-t administered during phone screening
* Able and willing to complete the 6 month protocol
* Not currently engaged in cognitive program
* No use of video games for more than 2 hours/week over the previous 2 years
* No plans to have travel outside of the US in the next 6 months

Additional criteria for MRI/sleep (in addition to the above criteria for EFIT):

* Willing to undergo an MRI of the brain two times during the EFIT study
* Be able to lie flat on the MRI table in a supine position for at least 60 minutes
* Pass the standard IRB-approved SELIC MRI-safety screening criteria (see MRI screen SELIC in CATS)
* Willing to use the study-provided Sleep Profiler for 2 nights twice during the study
* Willing to wear a study-provided FitBit throughout the study
* No pregnant or breast feeding
* Must be right handed
* Must have sufficient vision to see ANT task without glasses
* No contraindication to MRI per standard MRI safety screening
* No persons with significant claustrophobia
* No open wound on the scalp or forehead
* No allergy to extended exposure to synthetic fabrics, such as polyester or rayon
* No head tremors or tics
* No persons currently using any of the following: opioids, stimulants, or recreational drugs
* No medication changes in the past 2 weeks in anxiety or depression medications
* No medication changes in the past 2 months for sleep disorders

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Useful Field of View (UFOV) test at 14 and 26 weeks | Baseline, Immediate Post-test at 14 weeks, and 3 month follow-up at 26 weeks
  This computerized assessment includes four subtests assessing processing speed, divided attention and selective attention scored in ms.
Change from Baseline Daily Everyday Cognitive Assessment (DECA) at 14 and 26 weeks | Baseline, Immediate Post-test at 14 weeks, and 3 month follow-up at 26 weeks
  This computerized task assesses everyday function across simulated everyday tasks of medical, nutrition, and problem solving tasks. Task accuracy and speed are recorded.
Change from Baseline iFunction at 14 and 26 weeks | Baseline, Immediate Post-test at 14 weeks, and 3 month follow-up at 26 weeks
  This computerized task assesses everyday function across simulated everyday tasks of medical, travel, and communication tasks. An overall score reflecting time and accuracy (i.e., efficiency index) is calculated to reflect performance across the ifunction subtests the proprietary software determines the score. Higher scores are better for efficiency index.

SECONDARY OUTCOMES:
Change from Baseline Objective sleep at 14 weeks | Baseline and Immediate Post-test at 14 weeks
  The sleep profiler monitor is a proprietary FDA approved ambulatory sleep EEG device designed for in-home sleep architecture monitoring. The Profiler will provide sleep spindle data in seconds, a pertinent sleep characteristic linked to memory and learning as well as computer brain training. Sleep spindles are an EEG hallmark of non-rapid eye movement (NREM) and are typically clinically classified as bursts of synchronous ~12-15 Hz neuronal firing in thalamocortical networks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No